CLINICAL TRIAL: NCT07093554
Title: Cilta-Talq Fusion Study: A Phase 1b Study of Talquetamab Bridging Therapy Followed by Ciltacabtagene Autoleucel in Patients With Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Othman S Akhtar, MBBS, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00055520
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Relapse Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Bispecific Antibody; CAR-T therapy; Refractory Multiple Myeloma; Relapse Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Talquetamab and Ciltacabtagene autoleucel (Experimental): Participants with relapsed and/or refractory multiple myeloma (RRMM) will be administered talquetamab as a bridging therapy during CAR T-cell manufacturing and then receive Ciltacabtagene autoleucel CAR T-cell infusion after which they will be followed up to six months.
  Interventions: Drug: Talquetamab; Drug: Ciltacabtagene Autoleucel

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered subcutaneously.
Drug: Ciltacabtagene Autoleucel — Ciltacabtagene Autoleucel will be administered intravenously.

SUMMARY:
This is a single-arm, open-label, phase 1b study evaluating the safety and feasibility of using talquetamab as bridging therapy prior to cilta-cel in patients with relapsed and refractory multiple myeloma (RRMM).

DETAILED DESCRIPTION:
This study will enroll patients with RRMM who have received at least one prior line of therapy and are eligible for both commercial talquetamab and cilta-cel. Patients will enroll prior to apheresis. Following apheresis, patients will receive one cycle of talquetamab therapy. An additional cycle of talquetamab will be allowed if manufacturing delays result in an expected lymphodepletion date > 4 weeks from the last full dose of talquetamab in Cycle 1. Following successful manufacturing, patients will receive lymphodepleting chemotherapy and cilta-cel infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Histologically confirmed diagnosis of multiple myeloma with evidence of progressive disease as defined by the IMWG criteria.
3. Have measurable disease, defined as:

   1. Serum M-protein level ≥ 1.0 g/dL, or
   2. Urine M-protein level ≥ 200 mg/24 hours, or
   3. In patients without a measurable M-protein, an involved light chain level ≥ 10 mg/dL and an abnormal free light chain ratio.
4. Patient had at least one prior line of therapy (PLOT), including a proteasome inhibitor (PI), an anti-CD38 antibody, and an immunomodulatory drug (IMID).
5. Patient meets the requirements for the use of talquetamab, as per the most recent FDA prescription information.
6. Patient plans to receive cilta-cel and meets the criteria for commercial use as per the most recent FDA prescription information.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at screening.
8. Have the following clinical laboratory values at screening:

   Adequate bone marrow function:

   Hemoglobin* ≥ 8.0 g/dL; Absolute Neutrophil Count* ≥ 1,000/mcL; Absolute Lymphocyte Count* ≥ 200/mcL; Platelets* ≥ 25,000/mm^3

   *Transfusion and growth factor support within 72 hours allowed.

   Adequate hepatic function:

   Total Bilirubin < 2 mg/dL; Aspartate aminotransferase (Serum Glutamic Oxaloacetic Transaminase)/Alanine Aminotransferase < 5 times institutional upper limit

   Adequate renal function:

   Creatinine Clearance ≥ 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
9. Female patients must meet one of the following:

   1. Postmenopausal for at least one year before the screening visit, or
   2. Surgically sterile, or
   3. If they are of childbearing potential:

   i. Agree to practice two effective methods of contraception from the time of signing of the informed consent form through three months after the last dose of the study drug, AND ii. Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or iii. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)
10. Male patients, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:

    1. Practice effective barrier contraception during the entire study treatment period and through 90 days after the last study drug dose, OR
    2. Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
    3. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
11. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Prior treatment:

   1. Adoptive T-cell therapy (e.g., CAR T-cell therapy) at any time prior to enrollment.
   2. Bispecific antibody, investigational or approved, irrespective of its target, at any time prior to enrollment.
   3. Use of talquetamab prior to enrollment.
   4. Any therapy targeting BCMA or GPRC5D, including but not limited to antibody-drug conjugates and/or monoclonal antibodies.
   5. Prior allogeneic stem cell transplant at any time.
   6. Autologous stem cell transplant within 2 months of date of enrollment.
   7. High-dose cytotoxic chemotherapy (e.g., DCEP, KD-PACE, D-PACE) within 28 days of the enrollment date.
   8. Cytotoxic chemotherapy, such as cyclophosphamide, within 14 days of the enrollment date .
   9. Treatment with a PI, IMID, anti-CD38 antibody, or venetoclax within 7 days of the enrollment date.
   10. A cumulative dexamethasone dose of ≥ 100 mg within 14 days of the enrollment date .
   11. Radiation therapy within 7 days of the enrollment date.
2. No ongoing Grade ≥ 3 non-hematological adverse events from prior therapy.
3. Active central nervous system (CNS) involvement.
4. Have plasma cell leukemia (PCL).
5. Have unmeasurable disease (oligosecretory or non-secretory myeloma).
6. Have concomitant AL amyloidosis.
7. Patients with severe cardiac disease.

   1. Active heart disease with New York Heart Association class III or IV congestive heart failure.
   2. History of myocardial infarction, unstable angina, placement of drug-eluting or metallic stent, coronary artery bypass graft in the last ≤ 6 months.
   3. Ejection fraction ≤ 40% on transthoracic echocardiography.
   4. Severe non-ischemic cardiomyopathy.
8. Patients with pulmonary dysfunction requiring continuous supplemental oxygen ≥ 2L/minute.
9. Any serious medical condition such as:

   1. Disabling neurological or psychiatric conditions, including altered mental status, dementia, or any condition that could preclude the use of high-dose steroids and/or accurate assessment of neurotoxicity.
   2. Any condition that could impair the ability of the subject to receive any of the study drugs.
10. Infections:

    1. No new uncontrolled clinically significant bacterial, viral or fungal infections.
    2. HIV-positive patients on combination antiretroviral therapy are not eligible.
11. Pregnant women are excluded from this study because talquetamab and cilta-cel have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with talquetamab, breastfeeding should be discontinued if the mother is treated with talquetamab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
The number of subjects without serious adverse events following Ciltacabtagene Autoleucel infusion through Day +30. | Day+30 post Ciltacabtagene Autoleucel infusion
  SAEs will be assessed using the NCI CTCAE v5.0 during bridging therapy and for 30 days following infusion. Immune-mediated toxicities will be graded and assessed using the American Society for Transplantation and Cellular Therapy (ASTCT) consensus grading systems. SAEs that meet the definition of the primary endpoint analysis will include:
  1. Any Grade 5 AE.
  2. Any Grade ≥ 4 non-hematological treatment-related AE.
  3. Cytokine release syndrome (Grade ≥ 3), immune-cell effector associated neurotoxicity syndrome (Grade ≥ 3) or immune effector cell-associated hemophagocytic lymphohistiocytosis-like syndrome (IEC-HS) of any grade.

CONTACTS AND LOCATIONS:
Overall Officials: Othman Akhtar, MBBS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No